CLINICAL TRIAL: NCT05954013
Title: Evaluating the Clinical and Cost-effectiveness of a Combined Person-centred Intervention of Advance Care Planning (ACP) and Care Coordination for People With Parkinson's Disease and Their Family Caregiver(s)
Brief Title: Advance Care Planning and Care Coordination for People With Parkinson's Disease
Acronym: PD_Pal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: University of Padova (Other); University of Ioannina (Other); University College, London (Other); Estonian Movement Disorders Society (Unknown); Paracelsus Medical University (Other); Philipps University Marburg (Other); Skane University Hospital (Other); Mediolanum Cardio Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 108177; NL8180 (Registry Identifier: Dutch Trial Register (NTR))
Record Dates: First submitted 2023-05-25; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2022-08

CONDITIONS: Parkinson Disease; Parkinsonism
Keywords: Advance Care Planning
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The participant and care provider (PD_Pal nurse) will not be blinded. The outcome assessor will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD_Pal intervention (Experimental): Participants with Parkinson's disease receive usual care from their established neurology and/or home care team + the PD_Pal intervention.
  Interventions: Behavioral: PD_Pal intervention
- Control group (No Intervention): Participants with Parkinson's disease receive usual care from their established neurology and/or home care team.

INTERVENTIONS:
Behavioral: PD_Pal intervention — The PD_Pal intervention will be delivered by a nurse that is specifically trained to deliver the PD_Pal intervention, i.e. the PD_Pal nurse. In the PD_Pal intervention, the patient, family caregiver and PD_Pal nurse complete four steps wherein they discuss and compose a: 1) Individual care plan; 2) Proactive care plan; 3) Quality of life and end-of-life plan and; 4) Coordination and revision plan. Together these steps lead to the Parkinson Support Plan. To facilitate patients in taking these steps, all patients receive a Parkinson Support Plan workbook. This workbook consists of information and questions aligned with the four steps. Patients can utilize this workbook before, during, or after the conversations with the PD_Pal nurse.
  Arms: PD_Pal intervention

SUMMARY:
Background: People with Parkinson's disease (PD), including parkinsonisms, experience complex motor and non-motor symptoms, which become more hindering in the advanced stages of PD. Advance care planning (ACP) enables individuals to define goals and preferences for future medical treatment and serves to ensure that people receive treatment and care that is in line with their preferences during serious chronic illness. The effectiveness of ACP for PD is currently unknown.

Methods: The investigators will evaluate the effectiveness of a multicenter, open-label randomized controlled trial, with a parallel group design in seven European countries (Austria, Estonia, Germany, Greece, Italy, Sweden and United Kingdom). The "PD_Pal intervention" comprises (1) several consultations with a trained nurse who will perform ACP conversations and support care coordination and (2) use of a patient-directed "Parkinson Support Plan-workbook". The intervention group will be compared to a care-as-usual group. Documented ACP-decisions in the medical records/patient's central file assessed at 6 months after baseline will be the primary endpoint. Secondary endpoints include patients' and family caregivers' quality of life, perceived care coordination, patients' symptom burden, and cost-effectiveness. Assessments will take place at baseline, 6 months after baseline and 12 months after baseline. In parallel, we will perform a process evaluation, to understand the feasibility of the intervention.

Hypothesis: The investigators hypothesize that the PD_Pal intervention will result in an increased number of participants with ACP documentation in the medical records/patient's central file, as compared to care-as-usual. Secondly, the investigators expect that, due to the PD_Pal intervention, patients and their FC will experience better care coordination, better quality of life, a reduced patient symptom burden and the FC will experience a reduction in caregiver burden.

ELIGIBILITY:
Inclusion criteria for people with Parkinson's disease:

* Capable to participate , meaning that the subject is able to:

  * understand information about the decision
  * remember that information
  * use that information to make a decision
  * communicate their decision by talking, using sign language or any other means
* Able to provide informed consent;
* Meeting the MDS clinical diagnostic criteria for PD, including Parkinsonisms;
* Hoehn & Yahr ≥ 3;
* Progressive deterioration in physical and/or cognitive function despite optimal therapy, according to the primary physician; and
* Availability of a family caregiver or informal caregiver.

Exclusion Criteria:

* Inability to communicate independently, with or without supportive communication tools; - Unable or unwilling to commit to study procedures;
* Presence of additional chronic medical illnesses which may require palliative services (e.g. metastatic cancer);
* Already receiving palliative care or hospice services;
* Already participating in a clinical study for palliative care.

Inclusion criteria for family caregivers (FCs):

* Identified by the patient as the person closest to them;
* Willing to provide written informed consent;
* Willing and able to complete questionnaires;
* Aging ≥ 18 years.

FC can only participate when the patient participates.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Advance care planning documentation in the medical records | 6 months after baseline; score range: 0-100; higher scores indicate higher percentages (though higher scores are not better per definition).
  Percentage of participants with documented advance care planning (ACP) preferences and wishes in the medical records at 6 months. Only participants who did not have documented ACP at baseline are included in this calculation.

SECONDARY OUTCOMES:
Advance care planning documentation in the medical records | 12 months after baseline; score range: 0-100; higher scores indicate higher percentages (though higher scores are not better per definition).
  Percentage of participants with documented advance care planning (ACP) preferences and wishes in the medical records at 12 months. Only participants who did not have documented ACP at baseline are included in the calculation.
Integrated Palliative Care Outcome Scale (IPOS) | 6 and 12 months after baseline; IPOS score range = 0-64; higher scores are worse
  Change from baseline in palliative phase symptom severity
Edmonton Symptom Assessment Scale for Parkinson's Disease (ESAS-PD) | 6 months after baseline; ESAS-PD score range = 0-140; higher scores are worse
  Change from baseline in disease specific symptoms
Beck Depression Inventory (BDI-I) | 6 months after baseline; BDI-I score range = 0-63; higher scores are worse
  Change from baseline in depression severity
Parkinson's Disease Questionnaire-39 (PDQ-39) | 6 and 12 months after baseline; PDQ-39 score range = 0-100; higher scores are worse
  Change from baseline in quality of life
EQ-5D-5L (patient) | 6 and 12 months after baseline; EQ-5D-5L score range = 11111-55555; higher scores are worse
  Change from baseline in self-rated health status in 5 domains
Self-rated health status (patient), on a 0-100 point VAS scale | 6 and 12 months after baseline; score range: 0-100; higher scores indicated better self-rated health status
  Change from baseline in self-rated health status
EQ-5D-5L (family caregiver) | 6 and 12 months after baseline; EQ-5D-5L score range = 11111-55555; higher scores are worse
  Change from baseline of caregiver's health status in 5 domains
Quality of life questionnaire for carers - PQoL Carer | 6 and 12 months after baseline; PQoL Carer score range = 0-100; higher scores are worse
  Change from baseline in burden experienced by family caregiver
Modified Nijmegen Continuity Questionnaire (mNCQ) | 6 and 12 months after baseline; mNCQ score range = 1-5; higher scores are worse
  Change from baseline in perceived care coordination
Short Assessment of Patient Satisfaction (SAPS) | 6 months after baseline; SAPS score range = 0-32; higher scores are worse
  Change from baseline in quality of care
Experienced involvement in decision making (CollaboRATE) | 6 months after baseline; CollaboRATE score range = 0-5; higher scores are worse
  Change from baseline in experienced involvement in decision making.
MDS Non-Motor Rating Scale (MDS-NMS) | 6 and 12 months after baseline; MDS-MMS score range = 0-832; higher scores are worse
  Change from baseline in non-motor symptom severity
Quality of Dying and Death questionnaire (QoDD), if applicable | 30 days after death of patient; QoDD score range = 0-100; lower scores are worse
  Quality of the dying process, experienced by family caregiver
Resource Utilization questionnaire (RUD) adapted for PD | 6 and 12 months after baseline; RUD score range not applicable
  Change from baseline in resource utilisation

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Antonini, MD, PhD, Principal Investigator — University of Padova
Locations (7):
- Paracelsus Medical University, Salzburg, Austria
- Estonian Movement Disorders Society, Tartu, Estonia
- Philipps University Marburg Medical Center, Marburg, Germany
- University of Ioannina, Ioannina, Greece
- University of Padova, Padua, Italy
- Skane University Hospital, Lund, Sweden
- University College, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No